CLINICAL TRIAL: NCT07131111
Title: Impact of Aortic Geometry on Vascular Remodeling After Stent Implantation in Coarctation of the Aorta
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina wadee fathy, Principal investigator, Assiut University
Other Study IDs: Vascular remodeling in COA
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Aortic Geometry; Vascular Remodeling; Coarctation of Aorta; Blood Pressure; Residual Stenosis; CT Aortography; CMR; Aortic Elasticity and Distensibility; Aortic Arch
MeSH Terms: conditions — Vascular Remodeling; Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COA patients
  Interventions: Radiation: CT aortography; Radiation: CMR
- Healthy controls
  Interventions: Radiation: CT aortography

INTERVENTIONS:
Radiation: CT aortography — Performed before and after stenting using a multidetector CT scanner (device model and parameters to be specified).
  Analysis will include:
  * Evaluation of aortic arch geometry (normal / gothic / crenel).
  * Measurement of residual stenosis at the site of coarctation.
  * Aortic diameter measurements at predefined anatomical levels:
  Ascending aorta (AA), Proximal descending thoracic aorta (PDA), At the level of the diaphragm (DA), Abdominal aorta (AbAo).
  - Aortic tortuosity. All CT data will be interpreted by two independent observers blinded to clinical outcomes
Radiation: CMR — CMR examinations will be performed using a commercially available 1.5 Tesla whole-body scanner (Ingenia, Philips Healthcare, release 4.1.3.0). In pediatric or uncooperative patients, free-breathing sequences were used when breath-holding was not feasible.
  Brachial blood pressure was measured in the right arm in the supine position immediately before image acquisition using automated oscillometric devices.
  Cine steady-state free precession (SSFP) sequences were obtained in multiple views including the short axis of the ascending aorta (AAO) and descending aorta (DAO), as well as the aortic root to evaluate aortic valve morphology (bicuspid vs tricuspid).
  Left ventricular (LV) and left atrial (LA) functional parameters were assessed by standard volumetric analysis. The following CMR-derived parameters were collected:
  Left ventricular ejection fraction (LVEF) Left ventricular strain Left ventricular mass index (LVMI) Left atrial volume Left atrial strain LV and LA strain were analyzed usi
  Groups: COA patients

SUMMARY:
This study aims to assess:

1. Aortic geometrical changes and their relationship to hypertension and cardiovascular events.
2. Aortic geometrical differences between healthy individuals and patients with repaired coarctation of the aorta.

DETAILED DESCRIPTION:
Coarctation of the aorta (CoA) is a congenital narrowing of the aortic lumen, accounting for 5-8% of congenital heart diseases, with an incidence of 1 in 3000-4000 live births . This narrowing leads to altered hemodynamics, including increased left ventricular afterload, systemic hypertension, and long-term vascular remodeling, which can persist even after anatomical correction .

Despite advances in interventions like stent implantation for native or recurrent CoA, many patients remain hypertensive post-procedure . This residual hypertension may not be purely mechanical but linked to persistent vascular dysfunction, abnormal aortic compliance, or inadequate aortic wall remodeling .

Aortic stiffness is now recognized as a key cardiovascular risk factor in CoA patients . Reduced elasticity contributes to high systolic blood pressure, increased cardiac workload, and late cardiovascular complications [7]. Moreover, abnormal aortic arch geometry-particularly the "gothic arch"-has been linked to impaired vascular function and unfavorable hemodynamics [13].

While cardiac magnetic resonance (CMR) is the standard for evaluating aortic stiffness and ventricular function , CT Aortography offers high-resolution images to assess aortic distensibility, luminal changes, and residual stenosis, especially post-stenting . When combined with blood pressure and ECG data, these insights can provide a fuller picture of outcomes .

This study investigates the relationship between post-stenting blood pressure and aortic geometry-including arch shape and residual stenosis-using CT Aortography in CoA patients. It also explores ECG changes as potential non-invasive markers of ventricular strain and hemodynamic stress ..

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 12 years.

Diagnosed with native or recurrent coarctation of the aorta.

Transcatheter systolic pressure gradient ≥ 20 mmHg.

Body weight ≥ 20 kg.

Availability of pre- and post-stenting CT aortography data.

Exclusion Criteria:

Patients with obstructive lesion of LVOT or aortic valve dysfunction greater than moderate (requiring surgical intervention)..

Patients with other causes of secondary hypertension.

Associated complex congenital heart defects (aside from simple septal defects and patent ductus arteriosus)

Genetic syndromes

Connective tissue disorder

History of surgery involving the aortic root or ascending aorta.

Incomplete imaging or missing data relevant to the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of two groups:
  1. Patients group: Individuals diagnosed with coarctation of the aorta (CoA) who have undergone successful stent implantation and will be evaluated six months post-stenting.
  2. Control group: Age- and sex-matched healthy volunteers with no history of cardiovascular or systemic diseases.
  All participants will undergo imaging and functional evaluation including CT aortography, cardiac MRI, 24-hour ambulatory blood pressure monitoring (ABPM), and ECG as part of the study protocol.
  The study will be conducted at [Assiut University Hospital / Orman Cardiology Center - modify as needed], and participants will be recruited from the cardiology outpatient clinics and imaging units.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline and 6 months post-stenting
  Difference in systolic blood pressure between baseline (pre-stenting) and 6 months post-stenting using standardized clinical sphygmomanometer.
  Unit of Measure: mmHg
Change in Diastolic Blood Pressure | Baseline and 6 months post-stenting
  Difference in diastolic blood pressure between baseline (pre-stenting) and 6 months post-stenting using standardized clinical sphygmomanometer.
  Unit of Measure: mmHg

SECONDARY OUTCOMES:
Aortic Arch Morphology Classification | Baseline (within hospital stay, up to 2 days)
  Classification of aortic arch morphology (normal, gothic, crenel) based on CT aortography.
  Unit of Measure: Categorical (normal/gothic/crenel)
Aortic Elasticity | Baseline and 6 months post-stenting
  Aortic elasticity calculated from CT aortography using (ΔA/A)/ΔP, where A is cross-sectional area and P is pulse pressure.
  Unit of Measure: mm²/mmHg
Aortic Distensibility | Baseline and 6 months post-stenting
  Aortic distensibility measured from CT aortography. Unit of Measure: mmHg-¹
Aortic Arch Angle | Baseline and 6 months post-stenting
  Aortic arch angle measured from CT aortography. Unit of Measure: degrees
Aortic Arch Curvature | Baseline and 6 months post-stenting
  Curvature of the aortic arch measured from CT aortography. Unit of Measure: cm-¹
Residual Stenosis | 6 months post-stenting
  Percentage of luminal narrowing remaining after stent implantation measured by CT angiography.
  Unit of Measure: %
Left Ventricular Ejection Fraction (LVEF) | Baseline and 6 months post-stenting
  Description: LVEF measured by cardiac MRI. Unit of Measure: %
LV Global Longitudinal Strain | Baseline and 6 months post-stenting
  LV global longitudinal strain measured by cardiac MRI. Unit of Measure: %
LV Mass Index (LVMI) | Baseline and 6 months post-stenting
  LV mass indexed to body surface area measured by cardiac MRI. Unit of Measure: g/m²
Left Atrial Volume Index (LAVI) | Baseline and 6 months post-stenting
  Description: Left atrial volume indexed to body surface area measured by cardiac MRI.
  Unit of Measure: mL/m²
QTc Dispersion | Baseline and 6 months post-stenting
  QTc dispersion measured from 12-lead ECG using Bazett's formula. Unit of Measure: milliseconds
Presence of Left Ventricular Hypertrophy on ECG | Baseline and 6 months post-stenting
  Detection of LV hypertrophy based on standard ECG voltage criteria. Unit of Measure: Categorical (present/absent)
Presence of Arrhythmia | Baseline and 6 months post-stenting
  Detection of arrhythmias using standard 12-lead ECG or Holter monitoring. Unit of Measure: Categorical (present/absent)

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Demitry Roshdy, Professor, Study Director — Faculty of medicine AssiutU university
Locations (1):
- Institutional Review Board (IRB) of Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shepherd B, Abbas A, McParland P, Fitzsimmons S, Shambrook J, Peebles C, Brown I, Harden S. MRI in adult patients with aortic coarctation: diagnosis and follow-up. Clin Radiol. 2015 Apr;70(4):433-45. doi: 10.1016/j.crad.2014.12.005. Epub 2015 Jan 3. PMID 25559379
- [Background] Toro-Salazar OH, Steinberger J, Thomas W, Rocchini AP, Carpenter B, Moller JH. Long-term follow-up of patients after coarctation of the aorta repair. Am J Cardiol. 2002 Mar 1;89(5):541-7. doi: 10.1016/s0002-9149(01)02293-7. PMID 11867038
- [Background] Parati G, Stergiou GS, Asmar R, Bilo G, de Leeuw P, Imai Y, Kario K, Lurbe E, Manolis A, Mengden T, O'Brien E, Ohkubo T, Padfield P, Palatini P, Pickering T, Redon J, Revera M, Ruilope LM, Shennan A, Staessen JA, Tisler A, Waeber B, Zanchetti A, Mancia G; ESH Working Group on Blood Pressure Monitoring. European Society of Hypertension guidelines for blood pressure monitoring at home: a summary report of the Second International Consensus Conference on Home Blood Pressure Monitoring. J Hypertens. 2008 Aug;26(8):1505-26. doi: 10.1097/HJH.0b013e328308da66. PMID 18622223
- [Background] Iriart X, Laik J, Cremer A, Martin C, Pillois X, Jalal Z, Roubertie F, Thambo JB. Predictive factors for residual hypertension following aortic coarctation stenting. J Clin Hypertens (Greenwich). 2019 Feb;21(2):291-298. doi: 10.1111/jch.13452. Epub 2018 Dec 25. PMID 30585428
- [Background] Pushparajah K, Duong P, Mathur S, Babu-Narayan S. EDUCATIONAL SERIES IN CONGENITAL HEART DISEASE: Cardiovascular MRI and CT in congenital heart disease. Echo Res Pract. 2019 Oct 1;6(4):R121-38. doi: 10.1530/ERP-19-0048. Online ahead of print. PMID 31730044
- [Background] Faganello G, Cioffi G, Rossini M, Ognibeni F, Giollo A, Fisicaro M, Russo G, Di Nora C, Doimo S, Tarantini L, Mazzone C, Cherubini A, D'Agata Mottolesi B, Pandullo C, Di Lenarda A, Sinagra G, Viapiana O. Are aortic coarctation and rheumatoid arthritis different models of aortic stiffness? Data from an echocardiographic study. Cardiovasc Ultrasound. 2018 Jun 26;16(1):9. doi: 10.1186/s12947-018-0126-y. PMID 29940971
- [Background] Agasthi P, Pujari SH, Tseng A, Graziano JN, Marcotte F, Majdalany D, Mookadam F, Hagler DJ, Arsanjani R. Management of adults with coarctation of aorta. World J Cardiol. 2020 May 26;12(5):167-191. doi: 10.4330/wjc.v12.i5.167. PMID 32547712
- [Background] Ou P, Mousseaux E, Celermajer DS, Pedroni E, Vouhe P, Sidi D, Bonnet D. Aortic arch shape deformation after coarctation surgery: effect on blood pressure response. J Thorac Cardiovasc Surg. 2006 Nov;132(5):1105-11. doi: 10.1016/j.jtcvs.2006.05.061. PMID 17059930
- [Background] Ou P, Bonnet D, Auriacombe L, Pedroni E, Balleux F, Sidi D, Mousseaux E. Late systemic hypertension and aortic arch geometry after successful repair of coarctation of the aorta. Eur Heart J. 2004 Oct;25(20):1853-9. doi: 10.1016/j.ehj.2004.07.021. PMID 15474701
- [Background] Vonder Muhll IF, Sehgal T, Paterson DI. The Adult With Repaired Coarctation: Need for Lifelong Surveillance. Can J Cardiol. 2016 Aug;32(8):1038.e11-5. doi: 10.1016/j.cjca.2015.12.036. Epub 2016 Jan 21. PMID 27084076